CLINICAL TRIAL: NCT04518449
Title: the Medial Border Along the Left Side of SMA Versus the Left Side of SMV in Laparoscopic D3 Lymphadenectomy for Right Colon Cancer, a Prospective Cohort Study
Brief Title: Medial Border of Laparoscopic D3 Lymphadenectomy for Right Colon Cancer
Status: Withdrawn | Type: Observational
Why Stopped: no funds
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Principal Investigator, Cai Zhenghao, Attending surgeon of gastrointestinal surgery，Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai Minimally Invasive Surgery Center
Other Study IDs: MISC- Medial border of D3
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SMA group: the medial border along the left side of superior mesenteric artery (SMA)
  Interventions: Procedure: medial border along the left side of SMA
- SMV group: the medial border along the left side of superior mesenteric vein (SMV)
  Interventions: Procedure: medial border along the left side of SMV

INTERVENTIONS:
Procedure: medial border along the left side of SMA — to place the medial border along the left side of SMA in laparoscopic D3 lymphadenectomy for right colon cancer
  Groups: SMA group
Procedure: medial border along the left side of SMV — to place the medial border along the left side of SMV in laparoscopic D3 lymphadenectomy for right colon cancer
  Groups: SMV group

SUMMARY:
This study investigats the gastrointestinal functional outcomes of laparoscopic D3 lymphadenectomy for right colon cancer with the medial border along the left side of superior mesenteric artery (SMA) versus the left side of superior mesenteric vein (SMV). This is a single center, prospective cohort study with a sample size of 264 patients. The primary endpoint is the incidence of diarrhea (evaluated using the Diarrhea Assessment Scale) one month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* American Society of Anesthesiologists (ASA) score I to III
* A biopsy proven histological diagnosis of colorectal carcinoma
* tumor located at right half of colon
* Undergoing laparoscopic right hemi-colectomy
* preoperative staging cT2-4aN0M0 or cTanyN+M0
* willing to participate and informed consent signed

Exclusion Criteria:

* Pregnant or lactating women
* Synchronous colorectal carcinoma
* History of colorectal cancer or other malignant tumors
* Clinical evidence of metastasis
* Preoperative staging cT1N0 or cT4bNany
* Emergency procedure

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: conlon cancer located at right hemi-colon
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
incidence of diarrhea | one month after surgery
  Diarrhea Assessment Scale: stool score ≥ 5

IPD SHARING:
Plan to Share IPD: Undecided